CLINICAL TRIAL: NCT04384887
Title: ''(COVID-19) and Anxiety and Depressive Symptoms in Pregnant Women"
Brief Title: "Investigation of the Relationship Between New Coronary Virus Disease (COVID-19) and Anxiety and Depressive Symptoms in Pregnant Women"
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Collaborators: Ayşegül Bestel (Unknown); İbrahim Polat (Unknown); Merve Aldıkaçtıoğlu Talmaç (Unknown)
Responsible Party: Principal Investigator, Pınar Yalcin bahat, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: beckcovid
Record Dates: First submitted 2020-05-11; First posted 2020-05-12 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-05

CONDITIONS: COVID; Anxiety; Depression, Postpartum
MeSH Terms: conditions — Anxiety Disorders; Depression, Postpartum

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: covid-19 positive pregnant women — It is planned to receive pregnant women who are admitted to the clinic or outpatient clinic and who are offered inpatient follow-up and treatment with the diagnosis of COVID-19.
  Pregnant women who do not have covid-19 disease as a control group and who do not have a comorbid disease at similar gestational week will be included in the study. As a control group, covid-19 pcr negative patients will be admitted to our clinic in the same period.
  Other Names: covid-19 negative pregnant women

SUMMARY:
In our study; Anxiety and depression levels, socio-demographic characteristics of the pregnant women who were admitted to our hospital between 25.04.2020-25.07.2020 and treated with the diagnosis of covid 19, and the change in anxiety and depression levelsWİTH Beck Depression and Anxiety Score after the disease regressed are planned.

(Beck depression scale contains 10 questions and a total of 1 to 100 points is obtained. High score indicates that depression and anxiety are high.) 0-16 points = mild depressive symptoms

17-29 points = moderate depressive symptoms

30-63 points = severe depressive symptoms

DETAILED DESCRIPTION:
The sociodemographic data form prepared by the researchers will be filled out by interviewing the patients who are willing to participate in the study. In addition, Beck Depression Scale, Beck Anxiety Scale, State and Trait Anxiety Scale will be given by the participants themselves. When the patients come to their first control after discharge, the scales specified will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* covid -19 pcr positive pregnant women
* no psychiatric diagnosis no use of psychiatric medicine

Exclusion Criteria:

Non-pregnant patients, A psychiatric diagnosis use of psychiatric medicine

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Pregnant women with a positive covid -19 pcr test between the ages of 18 and 45 will be included in the study and beck and anxiety tests will be performed 3 months after birth.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-04-25 (Actual); Primary Completion 2020-08-25 (Actual); Study Completion 2020-08-26 (Actual)

PRIMARY OUTCOMES:
Evaluation of depression and anxiety score changes of covid-19 positive pregnants | 4 months
  Evaluation of depression and anxiety score changes of covid-19 positive pregnants Pregnant women are questioned how this period was affected, as the pandemic period loaded with extra stress and caused depression and anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Pinar Yalcin Bahat, Istanbul, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes